CLINICAL TRIAL: NCT05235360
Title: Factorial Trial to Test Unique and Combined Effects of Guided Thinking Tasks to Optimize a Physical Activity Intervention Among Underactive Adults
Brief Title: Factorial Trial Testing Guided Thinking Tasks to Optimize a Physical Activity Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Methodist University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Kansas Medical Center (Other); University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H21-003-BALA; R21CA260360 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-02-11 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): 1) Episodic future thinking; 2) Positive affect imagery; 3) Action planning; 4) High intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Positive affect imagery; Behavioral: Action planning; Behavioral: High dose
- Condition 2 (Experimental): 1) Episodic future thinking; 2) Positive affect imagery; 3) Action planning; 4) Low intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Positive affect imagery; Behavioral: Action planning; Behavioral: Low dose
- Condition 3 (Experimental): 1) Episodic future thinking; 2) Positive affect imagery; 3) High intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Positive affect imagery; Behavioral: High dose
- Condition 4 (Experimental): 1) Episodic future thinking; 2) Positive affect imagery; 3) Low intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Positive affect imagery; Behavioral: Low dose
- Condition 5 (Experimental): 1) Recent thinking; 2) Positive affect imagery; 3) Action planning; 4) High intervention dose
  Interventions: Behavioral: Positive affect imagery; Behavioral: Action planning; Behavioral: High dose; Behavioral: Recent thinking
- Condition 6 (Experimental): 1) Recent thinking; 2) Positive affect imagery; 3) Action planning; 4) Low intervention dose
  Interventions: Behavioral: Positive affect imagery; Behavioral: Action planning; Behavioral: Recent thinking; Behavioral: Low dose
- Condition 7 (Experimental): 1) Recent thinking; 2) Positive affect imagery; 3) High intervention dose
  Interventions: Behavioral: Positive affect imagery; Behavioral: High dose; Behavioral: Recent thinking
- Condition 8 (Experimental): 1) Recent thinking; 2) Positive affect imagery; 3) Low intervention dose
  Interventions: Behavioral: Positive affect imagery; Behavioral: Recent thinking; Behavioral: Low dose
- Condition 9 (Experimental): 1) Episodic future thinking; 2) Neutral imagery; 3) Action planning; 4) High intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Action planning; Behavioral: High dose; Behavioral: Neutral imagery
- Condition 10 (Experimental): 1) Episodic future thinking; 2) Neutral imagery; 3) Action planning; 4) Low intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Action planning; Behavioral: Neutral imagery; Behavioral: Low dose
- Condition 11 (Experimental): 1) Episodic future thinking; 2) Neutral imagery; 3) High intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: High dose; Behavioral: Neutral imagery
- Condition 12 (Experimental): 1) Episodic future thinking; 2) Neutral imagery; 3) Low intervention dose
  Interventions: Behavioral: Episodic future thinking; Behavioral: Neutral imagery; Behavioral: Low dose
- Condition 13 (Experimental): 1) Recent thinking; 2) Neutral imagery; 3) Action planning; 4) High intervention dose
  Interventions: Behavioral: Action planning; Behavioral: High dose; Behavioral: Recent thinking; Behavioral: Neutral imagery
- Condition 14 (Experimental): 1) Recent thinking; 2) Neutral imagery; 3) Action planning; 4) Low intervention dose
  Interventions: Behavioral: Action planning; Behavioral: Recent thinking; Behavioral: Neutral imagery; Behavioral: Low dose
- Condition 15 (Experimental): 1) Recent thinking; 2) Neutral imagery; 3) High intervention dose
  Interventions: Behavioral: High dose; Behavioral: Recent thinking; Behavioral: Neutral imagery
- Condition 16 (Experimental): 1) Recent thinking; 2) Neutral imagery; 3) Low intervention dose
  Interventions: Behavioral: Recent thinking; Behavioral: Neutral imagery; Behavioral: Low dose

INTERVENTIONS:
Behavioral: Episodic future thinking — Participants will listen to a guided thinking task directing them to think about themselves at a future, positive event and to imagine the event in vivid and specific detail.
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 2; Condition 3; Condition 4; Condition 9
Behavioral: Positive affect imagery — Participants will listen to a guided thinking task directing them to think about positive feelings and associations about physical activity in specific, personal, and positive detail.
  Arms: Condition 1; Condition 2; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Action planning — Participants will listen to a guided thinking task directing them to think about the remainder of their week and when, where, and how they plan to attain their remaining activity for the week.
  Arms: Condition 1; Condition 10; Condition 13; Condition 14; Condition 2; Condition 5; Condition 6; Condition 9
Behavioral: High dose — Participants will listen to the audio-recording with the guided thinking tasks 5 times/week.
  Arms: Condition 1; Condition 11; Condition 13; Condition 15; Condition 3; Condition 5; Condition 7; Condition 9
Behavioral: Recent thinking — Participants will listen to a guided thinking task directing them to think about a regular habit or activity they completed in the past week and to imagine that activity in specific and vivid detail.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Neutral imagery — Participants will listen to a guided thinking task directing them to imagine physical sensations (i.e., movements, muscles used) of a routine, daily activity (non-physical activity).
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Low dose — Participants will listen to the audio-recording with the guided thinking tasks 1 time/week.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The objective of this study is to optimize a novel, audio-recorded physical activity intervention that is scalable. Using principles of the Multiphase Optimization Strategy (MOST) framework, a full factorial study will test the unique and combined effects of different intervention components to identify which combination of components is optimal for increasing physical activity and mechanisms by which the components are or are not effective. This information will inform decisions about an optimal intervention package that is effective, efficient, and minimizes participant burden.

DETAILED DESCRIPTION:
Eligible participants who provide informed consent will be enrolled in a 6-week study. At the baseline session, participants will be randomized to listen to a brief audio-recording of different guided thinking tasks. The audio-recordings are based on combinations of four different intervention components that will be tested in a 2 (positive affect imagery vs. neutral) x 2 (episodic future thinking vs. recent thinking) x 2 (action planning: yes, no) x 2 (dose: high vs. low) factorial trial. Participants will also complete a 30-minute brisk walking session on a treadmill. Participants will return for weekly visits in which they again listen to their assigned audio-recording and complete a 30-minute brisk walking session.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-64
* Not currently meeting physical activity guidelines (<150 minutes/week of self-reported moderate-to-vigorous physical activity)
* Capable of providing informed consent
* Access to a smartphone with active data plan
* Willing to attend all study visits and comply with the protocol
* Conversant in English

Exclusion Criteria:

* BMI > 40
* orthopedic problems that would limit physical activity
* self-reported coronary artery disease, stroke, COPD, chronic bronchitis, emphysema, diabetes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in Weekly Physical Activity Minutes Across 6 Weeks (accelerometer-assessed) | Assessed weekly at Weeks 1-6
  Amount of weekly moderate-to-vigorous (MVPA) minutes (i.e., minutes of MPVA weighted by intensity) will be determined from accelerometers (ActiGraph wGT3X-BT) worn for one-week periods for six consecutive weeks.

SECONDARY OUTCOMES:
Change in Weekly Physical Activity Minutes Across 6 Weeks (self-reported) | Assessed weekly at baseline and at Weeks 1-6
  Amount of weekly self-reported MVPA (i.e., minutes of MPVA weighted by intensity) will be determined using the 7-day Physical Activity Recall (PAR) interview.

OTHER OUTCOMES:
Affective Response to Exercise | Assessed weekly at baseline and at Weeks 1-6
  The Feeling Scale measures affective responses to exercise on a -5 to +5 scale with higher scores indicated a more positive affective response. It will be assessed during- and post-exercise for the in-person brisk walking sessions. Will be assessed as a putative mechanism.
Intrinsic Motivation for Exercise | Assessed weekly at baseline and at Weeks 1-6
  The intrinsic subscale of the Behavioral Regulations in Exercise Questionnaire measures intrinsic motivation using a 0 to 4 response scale with higher scores indicating greater intrinsic motivation. It will be assessed after listening to the audio-recording in-person (post-intervention). Will be assessed as a putative mechanism.
Delayed Discounting | Assessed weekly at baseline and at Weeks 1-6
  The rapid delay discounting task will be assessed after listening to the audio-recording in-person (post-intervention). Will be assessed as a putative mechanism.
Action Planning | Assessed weekly at baseline and at Weeks 1-6
  The action planning scale (Sniehotta et al., 2005) measures action planning for physical activity on a 1 to 4 scale with higher scores indicating higher levels of planning. It will be assessed after listening to the audio-recording in-person (post-intervention). Will be assessed as a putative mechanism.
Physical Activity Intentions | Assessed weekly at baseline and at Weeks 1-6
  The physical activity intentions scale (Conner et al., 2017) measures intentions for physical activity on a 1 to 5 scale with higher scores indicating stronger intentions. It will be assessed after the in-person brisk walking session. Will be assessed as a putative mechanism.

CONTACTS AND LOCATIONS:
Overall Officials: Austin S. Baldwin, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available, in addition to the study protocol, statistical analysis plan, informed consent, and analytic code. Data will be made available to interested parties after all the initial study analyses and outcomes have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available one year after study completion.
Access Criteria: Researchers who provide a methodologically sound proposal and sign a data use agreement. Proposals should be submitted to Austin Baldwin.

REFERENCES:
- [Derived] Baldwin AS, Lamb CL, Geary BA, Mitchell AD, Kouros CD, Levens S, Martin LE. Testing and Optimizing Guided Thinking Tasks to Promote Physical Activity: Protocol for a Randomized Factorial Trial. JMIR Res Protoc. 2022 Sep 8;11(9):e40908. doi: 10.2196/40908. PMID 36074550